CLINICAL TRIAL: NCT06010550
Title: Validating a Clinical Decision Support Tool for Stratifying Stroke Risk in Patients Presenting With Dizziness to the Emergency Department
Brief Title: Validating a Clinical Decision Support Tool for Stratifying Stroke Risk for Dizziness/Vertigo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chiayi Christian Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB2023009
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Dizziness; Vertigo
Keywords: Dizzy; Vertigo; Stroke; Machine learning
MeSH Terms: conditions — Dizziness; Vertigo; Stroke | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dizziness/vertigo: Patients aged 20 or above, presenting to the emergency department with dizziness or vertigo.
  Interventions: Radiation: Magnetic resonance imaging

INTERVENTIONS:
Radiation: Magnetic resonance imaging — Brain magnetic resonance imaging

SUMMARY:
This study aims to validate a machine learning model that stratifies the risk of stroke in patients who present to the emergency department with dizziness or vertigo.

DETAILED DESCRIPTION:
This is a cross-sectional, hospital-based study, with no randomization procedure. Over a 21-month period, approximately 600 subjects will be enrolled. The study will assess the risk of stroke in each patient using a machine-learning model. To detect ischemic or hemorrhagic stroke, each patient will undergo a non-contrast brain magnetic resonance imaging study. The predictive performance of the machine-learning model will be evaluated in terms of accuracy, precision, recall, F1 score, and area under the receiver operating characteristics curve.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the emergency department with dizziness or vertigo
* Aged ≥ 20
* Dizziness or vertigo lasting for at least 1 hour and < 7 days
* Persistent dizziness or vertigo at the time of the examination at the emergency department

Exclusion Criteria:

* Having 5 or more prior episodes similar in quality, intensity, and duration to the current symptoms, with at least one episode more than a year prior and one within the past year
* Having frank stroke-like symptoms or signs, such as hemiparesis, facial asymmetry, dysarthria, dysphasia, ataxia, gaze palsy
* Consciousness disturbance, Glasgow coma scale < 13
* Severe dementia
* Recent stroke within 3 months
* Dizziness or vertigo thought to be the result of head injury, hypotension, medication/drug intoxication, hypoglycemia, electrolyte imbalance, anemia, hepatic encephalopathy, hydrocephalus, etc
* Concomitant head or neck trauma
* Severe degenerative cervical spondylosis
* Having contraindications to magnetic resonance imaging examination

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who visit the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with stroke | Between 24 hours and 14 days after the emergency department visit
  Number of participants with ischemic or hemorrhagic stroke confirmed by brain magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Feng Sung, MD, PhD, Principal Investigator — Ditmanson Medical Foundation Chia-Yi Christian Hospital

IPD SHARING:
Plan to Share IPD: Undecided